CLINICAL TRIAL: NCT01117662
Title: Efficacy of Rituximab in Acute Cellular Rejection With B-cell Infiltrates in Renal Transplant Patients - Randomized Placebo Controlled Double Blind Trial
Brief Title: Efficacy of Rituximab in Acute Cellular Rejection in Renal Transplant Patients
Acronym: RIACT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The planned recruitment number of 180 Patient could not been achieved.
Sponsor: Hannover Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200710602
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Acute Rejection
Keywords: transplantation; acute rejection; kidney
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Intravenous application of Rituximab 375mg/m² body surface in 250 ml NaCl 0,9 % over 4 hours
  Interventions: Drug: Rituximab
- Control (Placebo Comparator): Intravenous application of placebo (NaCl 0,9 %) matching active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Intravenous application of Rituximab 375mg/m² body surface in 250 ml NaCl 0,9 % over 4 hours
  Other Names: MabThera
  Arms: Rituximab
Drug: Placebo — Intravenous application of placebo (NaCl 0,9 %) matching active treatment
  Arms: Control

SUMMARY:
Acute kidney allograft rejection is the major cause for a loss of graft function and has a negative impact on long-term graft survival. Anti-rejection therapy traditionally focuses on T cell-mediated mechanisms of renal allograft rejection. However, available agents that affect T-cell pathways have only little impact on long-term graft survival. There is increasing evidence that B-cells play an important role in acute transplant rejections. CD20+ B cell infiltrates in acute T-cell mediated rejections are frequent and correlate with a worse response to conventional anti-rejection treatment and an increased risk of graft loss. In one pilot study, supported by several case reports, a beneficial effect of Rituximab for the treatment of acute rejection episodes with intrarenal B-cell infiltrates was shown. However, despite the promise of these observations solid evidence is required before incorporating this treatment option into a general treatment recommendation.

In a multicenter randomized placebo controlled double blind phase III trial the investigators want to demonstrate that Rituximab in addition to standard treatment with steroid-boli is superior to the standard treatment alone regarding long-term kidney function. If the proposed study proves that Rituximab treatment of acute rejections is beneficial for the long-term allograft function, the conventional rejection therapy needs to be revised to this novel concept of B- cell targeting

ELIGIBILITY:
Inclusion criteria:

1. male or female patients age ≥ 18 at the time of the inclusion in the study
2. male or female patients after kidney transplantation if medically justifiable (cave: previous immunosuppression, particularly prior induction therapies or biologicals).
3. Proof of an acute rejection in kidney transplant according to Banff-criteria: T-cell-mediated rejection as borderline, grade IA/B, IIA/B (no v-only), if one or more results are available as significant B-cell infiltrates CD20≥20 / high power field, glomerulitis, peritubular capillaritis or C4d positivity (with the exception of ABO-incompatible transplantations) as well as patients who have no T-cell-mediated acute rejection, but signs of acute humoral rejection (as listed above according to the criteria glomerulitis, peritubular capillaritis, C4d positivity) who have to be treated according to medical opinion of the physician with steroid therapy. The evidence of rejection can be performed by a protocol or indication biopsy.
4. SV40-negativity in the biopsy
5. GFR calculated using the MDRD-Formula > 25 ml/min/1,73 m² in the time period before the noticed rejection.
6. Presence of a negative pregnancy test and consent to a highly effective contraceptive method (i.e. failure rate less than 1% per year, which are implants, injectable contraceptives, combined oral contraceptives, intrauterine devices (only hormone spirals), sexual abstinence or vasectomy of the partner) in patients of child-bearing age. This is not required when bilateral sterilization or ovariectomy of the patient and in patients that have exclusively female sex partners. Presence of consent to a highly effective contraceptive method for male patient.
7. Informed consent

Exclusion criteria:

1. Known contraindications, resp. incompatibility for Rituximab and/or for the concomitant medication
2. Administration of Rituximab within the last 12 months before inclusion
3. Simultaneous participation in an other clinical study or participation in an other clinical study within the last 30 days
4. Breastfeeding women or pregnant women
5. Persons who fail to assess essence, meaning and significance of the clinical study and act along these lines (according to § 40 Abs. 4 and § 41 Abs. 2 and Abs. 3 AMG)
6. Existence of an active CMV-infection, existence of a HIV-infection, existence of a replicative hepatitis B or C, existence of other grave infections
7. Cardiac insufficiency in phase NYHA III-IV
8. High grade cardiac arrhythmias
9. Unstable coronary heart disease
10. Poorly adjusted diabetes mellitus (HbA1c > 10 %) at the time of the inclusion in the study.
11. State after splenectomy
12. Contra-indication referring to a renewed transplant biopsy (e.g. coagulopathy, anticoagulation)
13. Other exclusion criteria according to the estimate of the attending doctor (e.g. aggravation of the general health condition, occurrence of a malignant disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Change of the GFR (glomerular filtration rate) one year after intervention compared to the baseline GFR before the rejection, which is calculated by a defined algorithm | Baseline, 1 year

SECONDARY OUTCOMES:
Progression of interstitial fibrosis and tubular atrophy between the biopsy that led to enrolment in the study and a scheduled protocol biopsy one year after intervention ("∆IFTA-Score") | 1 year

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (14):
  - Hannover Medical School, Hanover, Lower Saxony
  - Universitätsklinikum der RWTH Aachen Medizinische Klinik II, Aachen
  - Charité Campus Mitte Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln Medizinische Klinik IV Nephrologie, Cologne
  - Kliniken der Stadt Köln gGmbH Medizinische Klinik I, Cologne
  - Universitätsklinikum Düsseldorf Klinik für Nephrologie, Düsseldorf
  - Universitätsklinikum Erlangen Nephrologie und Hypertensiologie, Erlangen
  - Universitätsklinikum Essen Klinik für Nephrologie, Essen
  - Universitätsklinikum Freiburg Medzinische Klinik IV Nephrologie Freiburg, Freiburg im Breisgau
  - Nephrologisches Zentrum Niedersachsen 34346 Hannoversch Münden, Hannoversch Münden
  - Universitätsklinikum Jena Klinik für Innere Medizin III, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Kiel Klinik für Nieren- und Hochdruckkrankheiten Kiel, Kiel
  - Medizinische Klinik und Poliklinik I der Ludwig-Maximilians-Uniklinik München Klinikum Großhadern, München
  - Universitätsklinikum Münster Innere Medizin / Nephrologie, Münster

REFERENCES:
- [Derived] Schiffer L, Schiffer M, Merkel S, Schwarz A, Mengel M, Jurgens C, Schroeder C, Zoerner AA, Pullmann K, Brocker V, Becker JU, Dammrich ME, Trader J, Grosshennig A, Biertz F, Haller H, Koch A, Gwinner W. Rationale and design of the RIACT-study: a multi-center placebo controlled double blind study to test the efficacy of RItuximab in Acute Cellular tubulointerstitial rejection with B-cell infiltrates in renal Transplant patients: study protocol for a randomized controlled trial. Trials. 2012 Oct 26;13:199. doi: 10.1186/1745-6215-13-199. PMID 23101480